CLINICAL TRIAL: NCT00543192
Title: Sexual Functioning in Endometrial Cancer Survivors
Brief Title: Sexual Functioning in Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: CC07703; H-2007-0204 (Other: Institutional Review Board); A532820 (Other: UW Madison); SMPH/OBSTET & GYNECOL (Other: UW Madison)
Record Dates: First submitted 2007-10-10; First posted 2007-10-12 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2009-09

CONDITIONS: Endometrial Cancer; Sexual Function
Keywords: Endometrial Cancer; Sexual Function
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is estimate how sexual function in endometrial cancer survivors varies with severity of disease.

ELIGIBILITY:
Inclusion Criteria:

* History of Stage I-IIIA endometrial adenocarcinoma of any grade
* 1-5 years out from primary surgical treatment
* Adjuvant therapy may only have consisted of radiation or hormonal therapy
* No evidence of disease

Exclusion Criteria:

* Previous treatment for other malignancies
* Did not undergo surgery for primary treatment of endometrial cancer
* Inability to read, write and speak fluent English
* Major cognitive impairment affecting ability to provide consent

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University of Wisconsin Gynecologic Oncology and Radiation Oncology Clinics
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2007-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Female Sexual Function Index (FSFI). | at time of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: David M Kushner, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

REFERENCES:
- [Result] Onujiogu N, Johnson T, Seo S, Mijal K, Rash J, Seaborne L, Rose S, Kushner DM. Survivors of endometrial cancer: who is at risk for sexual dysfunction? Gynecol Oncol. 2011 Nov;123(2):356-9. doi: 10.1016/j.ygyno.2011.07.035. PMID 21855974
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu